CLINICAL TRIAL: NCT06488534
Title: The Effect of Intracolonic Infusion of FODMAPS on Colonic Motility and Symptoms in Healthy Volunteers
Brief Title: Intracolonic FODMAP Infusion in Healthy Volunteers
Acronym: ICOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University of Auckland, New Zealand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: S67510
Record Dates: First submitted 2023-09-12; First posted 2024-07-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2024-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — polyol

STUDY DESIGN:
Intervention Model Description: Mannitol, fructans and fructose will be intracolonically administered on 3 different intervestigation days with at least 2 weeks between each investigation day to avoid overlap of the different FODMAPs and to allow the colon to return to its original state
Who Masked: Participant, Investigator
Masking Description: Both the investigator and the participants will be blinded, which means that they will not know which of the 3 FODMAPs is administered
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fructose (Other): A solution of 10 g fructose in 200 mL of tap water will be infused once over a period of 20min. during 1 of the 3 investigation days.
  Interventions: Dietary Supplement: Fermentable Oligo-, Di- Monosaccharides And Polyols (FODMAPs)
- Fructan (Other): A solution of 30 g fructan in 200 mL of tap water will be infused once over a period of 20min. during 1 of the 3 investigation days.
  Interventions: Dietary Supplement: Fermentable Oligo-, Di- Monosaccharides And Polyols (FODMAPs)
- Mannitol (Other): A solution of 10 g mannitol in 200 mL of tap water will be infused once over a period of 20min. during 1 of the 3 investigation days.
  Interventions: Dietary Supplement: Fermentable Oligo-, Di- Monosaccharides And Polyols (FODMAPs)

INTERVENTIONS:
Dietary Supplement: Fermentable Oligo-, Di- Monosaccharides And Polyols (FODMAPs) — A FODMAP solution of 200 mL will be infused in the colon for over 20 min. via the lumen of the solid-state catheter for high-resolution colonic manometry.

SUMMARY:
Irritable bowel syndrome (IBS) is one of the most common chronic diseases of the gut-brain axis. The underlying pathophysiology is multifactorial, poorly understood and differs between the subtypes: constipation-dominant IBS, diarrhea-dominant IBS, mixed IBS, and unspecified IBS. Although it is considered a motility disorder, no uniform motility patterns have been found in IBS patients and no link has yet been found between the motility patterns and the typical complaints such as nausea, fullness, cramps and flatulence. These symptoms are often diagnosed after a meal and research has shown that especially fermentable oligo, di, monosaccharides and polyols (FODMAPs) give rise to symptoms. Many studies have tested the effect of these FODMAPs after oral administration, but little is known about their direct effect on the colon. In this double-blind cross-over study, 15 healthy volunteers are subjected to 3 colonoscopies in which a catheter is placed to measure the pressures in the large intestine and to administer the dissolved FODMAPs. Volunteers will follow a diet low in fiber and FODMAPs 3 days before each study visit. In addition, they will have to record their daily bowel movements during the week of their study visit and fill in 2 short questionnaires on the day of the study visit regarding their gastrointestinal complaints. There will be at least 2 weeks between the 3 study visits to avoid any overlap between the FODMAPs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should provide written informed consent to participate in the study
* Women of child-bearing potential agree to apply a highly effective method of birth control during the entire duration of the trial. Highly effective birth control is defined as those which result in a low failure rate (i.e., less than 1% per year) when used constantly and correctly such as implants, injectables, combined oral contraceptive method, or some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. Women of non-childbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or postmenopausal with at least 2 years without spontaneous menses.
* Subjects who are capable to understand the study and the questionnaires, and to comply with the study requirements.
* Healthy volunteers should consider themselves healthy and should not be medically examined

Exclusion Criteria:

* History of major surgery of the gastrointestinal tract (appendectomy, hemorrhoidectomy, or polypectomy greater than 3 months post-surgery are allowed).
* Known underlying organic gastrointestinal disease, including intestinal obstruction, ileus, intestinal perforation, severe inflammatory disorder like ulcerative colitis, Crohn's disease or toxic megacolon
* Diabetes mellitus types 1 and 2
* Concomitant Kidney or Liver disease, Biliary obstruction
* Decreased cardiac -or respiratory function
* Pregnant or breastfeeding women
* Use of antibiotics in the past month
* History of skin allergies or a history of extreme sensitivity to cosmetics or lotions
* Fragile skin vulnerable to skin tears.
* Damaged epigastric skin (open wounds, rash, inflammation)
* Subjects who are unable to remain in a relaxed reclined position for the test duration
* Subject has received an investigational drug or used an investigational medical device within 30 days prior to randomization, or is currently enrolled in an investigational study.
* The use of following drugs 1 month prior to inclusion and during the whole study duration: laxatives, opioids, anti-acids, anticholinergics/antispasmodics, anticonvulsants, antidepressants, diuretics, antihypertensives, antipsychotics, calcium channel blockers, bile acid sequestrants, iron supplements, anticoagulants, HIV protease inhibitors (saquinavir, lopinavir), atorvastatine, negazodone, efavirenz, Sint-janskruid (CYP3A4 inducers)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
colonic motility | through study completion, an average of 1 year
  evaluation of (high amplitude) propagating contractions, simultaneous pressure waves at 3 predefined timepoints: upon awakening, after FODMAP infusion and postprandially

SECONDARY OUTCOMES:
abdominal symptoms | through study completion, an average of 1 year
  symptoms will be registered every 15minutes during the evaluation of the colonic motility
stool form based on the bristol stool chart | through study completion, an average of 1 year
  stool form differences will be evaluated during the week of the investigation (3 days before the study visit, on the day of investigation, and 3 days after the study visit)
IBS-SSS and IBS-Qol | through study completion, an average of 1 year
  IBS symptom severity and influence of quality of life will be assessed at each investigation and compared between the 3 study arms.
microbiome | through study completion, an average of 1 year
  a stool sample will be taken before the first study visit to evaluate the microbial composition
colonic motor patterns by means of high resolution electrocolonography | through study completion, an average of 1 year
  simultaneous evaluation of colonic motor patterns with high-resolution colonic manometry and high-resolution electrocolonography
validation of the high-resolution electrocolonography | through study completion, an average of 1 year
  evaluation of the high-resolution electronography als a non-invasive tool for the measurement of colonic motility

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium